CLINICAL TRIAL: NCT04020250
Title: Echocardiographic Parameters in Predicting Outcome in Patients With Intermediate - Risk Pulmonary Embolism
Brief Title: Role of Echocardiography in Pulmonary Embolism
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rofaida Raafat Talaat Ibrahim, Principle Investigator, Assiut University
Other Study IDs: Echo in Pulmonary Embolism
Record Dates: First submitted 2019-07-09; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Echocardiography — Echocardiographic parameters:
  Tricuspid annulus plane systolic excursion (TAPSE) Tricuspid regurgitation peak gradient (TRPG)

SUMMARY:
1. To analyze the diagnostic and prognostic value of echocardiographic parameters.
2. Prediction of APE-related 30-day mortality and adverse out comes.
3. The need for rescue thrombolysis in initially normotensive Acute pulmonary embolism (APE) patients.

DETAILED DESCRIPTION:
Acute pulmonary embolism (APE) is the most serious clinical presentation of venous thromboembolism (VTE). According to registries and hospital discharge databases of unselected patients with Acute pulmonary embolism and venous thromboembolism , 30-day all-cause mortality rates are between 9% and 10%.

According to the recent European Society of Cardiology (ESC) guidelines on the diagnosis and treatment of Acute pulmonary embolism patients, clinical classification of the severity of an episode of Acute pulmonary embolism is based on the estimated 30-day Acute pulmonary embolism - related mortality risk. Patients with cardiogenic shock caused by Acute pulmonary embolism comprise a high-risk group for early death, which is estimated at more than 15%.

Fortunately most Acute pulmonary embolism patients are hemodynamically stable at admission but the early mortality risk is different in this population. Risk stratification of non-high-risk Acute pulmonary embolism patients is based on clinical presentation, cardiac laboratory biomarkers, and signs of right ventricular (RV) dysfunction on echocardiography or computed tomography. Low-risk patients require a short hospital stay and can be early discharged home or even treated as outpatients.

Intermediate-risk subjects comprise a very heterogeneous group in which the early mortality ranges between 2% and 15%. More of these patients stabilize hemodynamically during anticoagulation, but in some of them clinical deterioration occurs and therefore they may require rescue thrombolysis or surgical or percutaneous embolectomy.

Echocardiography is a useful diagnostic tool to detected right ventricular (RV) dysfunction. It was reported that tricuspid annulus plane systolic excursion (TAPSE) can be used for risk stratification of normotensive APE patients. The tricuspid regurgitation peak gradient (TRPG) is an echocardiographic sign of RV overload and it can also be used for risk stratification in Acute pulmonary embolism .

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 and <70 years.
2. Patients with intermediate- risk pulmonary embolism will be

   1. -hemodynamically stable at admission with systolic blood pressure

      * 90 mmHg and without signs of peripheral hypoperfusion.
   2. - elevated cardiac biomarkers levels (particularly, a positive cardiac troponin test

Exclusion Criteria:

* 1- Age <18 years.

  2- Patients diagnosed with chronic thromboembolic hypertension.

  3- Patients with valvular heart diseases.

  4- Patients with lung cancer.

  5- Acute massive pulmonary embolism.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with pulmonary embolism confirmed by contrast-enhanced multidetector computed tomography (MDCT) when thrombo-emboli were visualized
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
the need for rescue thrombolysis in initially normotensive Acute pulmonary embolism patients. | one month
  analyses the diagnostic and prognostic value of a new echocardiographic parameter, TRPG/ TAPSE, for prediction of APE-related 30-day death or the need for rescue thrombolysis in initially normotensive Acute pulmonary embolism patients.

REFERENCES:
- [Background] Bernard S, Namasivayam M, Dudzinski DM. Reflections on Echocardiography in Pulmonary Embolism-Literally and Figuratively. J Am Soc Echocardiogr. 2019 Jul;32(7):807-810. doi: 10.1016/j.echo.2019.05.007. No abstract available. PMID 31272591
- [Background] Kanar BG, Sahin A, Gol G, Ogur E, Kavas M, Atas H, Mutlu B. Timing and magnitude of regional right ventricular function and their relationship with early hospital mortality in patients with acute pulmonary embolism. Anatol J Cardiol. 2019 Jun;22(1):26-32. doi: 10.14744/AnatolJCardiol.2019.38906. PMID 31264657
- [Background] Kanar BG, Gol G, Ogur E, Kavas M, Atas H, Mutlu B. Assessment of right ventricular function and relation to mortality after acute pulmonary embolism: A speckle tracking echocardiography-based study. Echocardiography. 2019 Jul;36(7):1298-1305. doi: 10.1111/echo.14398. Epub 2019 Jun 11. PMID 31184782